CLINICAL TRIAL: NCT03093974
Title: Double-blind, Placebo-controlled, Clinical Trial on Efficacy and Safety of 12-months Therapy With Inhaled Colistimethate Sodium in the Treatment of Subjects With Non-cystic Fibrosis Bronchiectasis Chronically Infected With P. Aeruginosa
Brief Title: Efficacy and Safety of Inhaled CMS in Bronchiectasis Subjects With Chronic P. Aeruginosa Infection. (PROMIS-I)
Acronym: PROMIS-I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zambon SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Z7224L01; 2015-002743-33 (EudraCT Number)
Record Dates: First submitted 2017-03-09; First posted 2017-03-28 (Actual); Results first posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-01

CONDITIONS: Non Cystic Fibrosis Bronchiectasis
Keywords: Colistimethate Sodium; CMS
MeSH Terms: interventions — colistinmethanesulfonic acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CMS (Colimesthate sodium) (Experimental): Inhaled colistimethate sodium twice daily. The active pharmaceutical ingredient consisting of pure CMS one million international units (MIU) / 80 mg of CMS / 33 mg colistin base activity (CBA) was provided as a powder for nebuliser solution in 10R International Organization for Standardization (ISO) glass vials.
  Interventions: Drug: CMS
- Placebo (Placebo Comparator): Saline solution inhaled twice daily, provided and administered at the same way of the IMP.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CMS — 1 MIU equivalent to 80 mg colistimethate sodium diluted in 1 mL saline solution 0.45%. Investigational Medicinal Product (IMP) glass vials were shrink wrapped in opaque white plastic and provided in boxes of 30 vials (two weeks of b.i.d dosing).
  The 1 MIU/mL CMS/0.45% saline solution was transferred from the glass vial into a specific nebuliser system fitted with a 0.3 mL medication chamber, for administration by inhalation. This delivered a nominal dose of 0.3 MIU/24 mg CMS (~10 mg CBA) from the device.
  The first dose of the IMP was administered at the site under the supervision of the site staff and subjects were instructed how to prepare and self-administer the IMP at home via a specific nebuliser system, b.i.d (morning and evening) over a period of 12 months.
  At least 10 minutes (min) before each administration, an inhaled short-acting bronchodilator (e.g., salbutamol /albuterol), supplied by the Sponsor, could be taken to improve tolerability.
  Other Names: Colistimethate Sodium
  Arms: CMS (Colimesthate sodium)
Other: Placebo — 1 ml saline solution 0.45%. the placebo was made up of identical empty glass vials to which the same saline diluent was added in exactly the same way as the reconstitution of the active treatment by injecting the diluent through the rubber stopper. The glass vials were shrink wrapped with opaque white plastic to maintain the blind.
  Other Names: Saline Solution
  Arms: Placebo

SUMMARY:
The objective of the trial was to investigate the effect of the use of inhaled CMS, administered b.i.d. via a specific nebuliser for 12 months, compared to placebo in subjects with NCFB chronically infected with P. aeruginosa on the annualised frequency of pulmonary exacerbations.

DETAILED DESCRIPTION:
This was a randomised, multi-centre, double-blind, placebo-controlled, parallel group interventional trial in subjects with NCFB and chronic P. aeruginosa infection. Subjects were randomised to CMS or placebo in a 1:1 ratio. The study consisted of seven clinic visits over one year with a follow-up phone call two weeks after discontinuation of treatment. Additional clinic visits, where feasible,and weekly phone calls were conducted during or after pulmonary exacerbations (or any episodes of pneumonia) until resolution.

All planned and unscheduled visits were preferably performed at sites, whenever possible. If on site visits after Visit 2 could not be performed at site due to COVID-19, remote visits (e.g., by telephone) were permitted. Mandatory on site visits were kept for Screening Visit (Visit 1) and Randomisation (Visit 2). If the final visit (Visit 7) had to be conducted remotely, then subjects were asked to return to the clinic for on-site assessments at the earliest opportunity.

ELIGIBILITY:
Inclusion Criteria:

1. are able and willing to give informed consent, following a detailed explanation of participation in the protocol and signed consent obtained;
2. aged 18 years or older of either gender;
3. diagnosed with NCFB by computerised tomography (CT) or high resolution CT (HRCT) as recorded in the subject's notes and this is their predominant condition being treated;
4. had at least 2 NCFB pulmonary exacerbations requiring oral or inhaled antibiotics or 1 NCFB pulmonary exacerbation requiring intravenous antibiotics in the 12 months preceding the Screening Visit (Visit 1) and had no NCFB pulmonary exacerbation with or without treatment during the period between Visit 1 and Visit 2;
5. have a documented history of P. aeruginosa infection ;
6. are clinically stable and have not required a change in pulmonary treatment for at least 30 days before the Screening Visit (Visit 1);
7. have pre-bronchodilator FEV1 ≥25% of predicted;
8. had a positive sputum culture for P. aeruginosa from an adequate sample taken at the Screening Visit (Visit 1) or during the screening period.

Exclusion Criteria:

1. known bronchiectasis as a consequence of cystic fibrosis (CF);
2. known history of hypogammaglobulinaemia requiring treatment with immunoglobulin, unless fully replaced and considered immuno-competent by the Investigator;
3. myasthenia gravis or porphyria;
4. severe cardiovascular disease such as severe uncontrolled hypertension, ischaemic heart disease or cardiac arrhythmia and any other conditions that would confound the evaluation of safety, in the opinion of the Investigator;
5. had major surgery in the 3 months prior to Screening Visit (Visit 1) or planned inpatient major surgery during the study period;
6. receiving treatment for allergic bronchopulmonary aspergillosis (ABPA);
7. had massive haemoptysis (greater than or equal to 300 mL or requiring blood transfusion) in the preceding 4 weeks before Screening Visit (Visit 1) or between Visit 1 and Visit 2;
8. respiratory failure that would compromise patient safety or confound the evaluation of safety or efficacy of the study in the opinion of the Investigator;
9. current active malignancy, except for basal cell carcinoma or squamous cell carcinoma of the skin without metastases;
10. taking immunosuppressive medications (such as azathioprine, cyclosporine, tacrolimus, sirolimus, mycophenolate, rituximab), and/or anti-cytokine medications (such as anti IL-6 and anti-tumour alpha necrosis factor products) in the preceding year before the Screening Visit (Visit 1);
11. known history of human immunodeficiency virus (HIV);
12. current treatment for non-tuberculous mycobacterial (NTM) lung disease or tuberculosis;
13. known or suspected to be allergic or unable to tolerate colistimethate sodium (intravenous or inhaled) or other polymixins, including previous evidence of bronchial hyperreactivity following inhaled colistimethate sodium;
14. treatment with long term (≥ 30 days) prednisone at a dose greater than 15 mg a day (or equivalent dose of any other corticosteroid) within six months of the Screening Visit (Visit 1)
15. new maintenance treatment with any oral macrolides (e.g. azithromycin/erythromycin/clarithromycin) started within 30 days of the Screening Visit (Visit 1) and between Visit 1 and Visit 2;
16. use of any intravenous or intramuscular or oral or inhaled antipseudomonal antibiotic (except chronic oral macrolide treatment with a stable dose) within 30 days prior to Screening Visit (Visit 1) and between Visit 1 and Visit 2;
17. pregnant or breast feeding or plan to become pregnant over the next year or of child bearing potential and unwilling to use a reliable method of contraception for at least one month before randomisation and throughout their involvement in the trial;
18. significant abnormality in clinical evaluations and/or laboratory tests (physical examination, vital signs, haematology, clinical chemistry, clinically relevant impaired renal function, defined as serum creatinine levels ≥2.0x upper limit of normal, ECG) endangering the safe participation of the patient in the study at the Screening Visit (Visit 1) and during the study;
19. participated in another investigational, interventional trial within 30 days prior to the Screening Visit (Visit 1);
20. in the opinion of the Investigator not suitable for inclusion for whatever reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (74):
- Australia (11):
  - Zambon Investigative Site, Adelaide
  - Zambon Investigative Site, Chermside
  - Zambon Investigative Site, Concord
  - Zambon Investigative Site, Frankston
  - Zambon Investigative Site, Greenslopes
  - Zambon Investigative Site, Melbourne
  - Zambon Investigative Site, Nedlands
  - Zambon Investigative Site, New Lambton Heights
  - Zambon Investigative Site, South Brisbane
  - Zambon Investigative Site, Spearwood
  - Zambon Investigative Site, Westmead
- Belgium (2):
  - Zambon Investigative Site, Ghent
  - Zambon Investigative Site, Roeselare
- Germany (8):
  - Zambon Investigative Site, Berlin
  - Zambon Investigative Site, Essen
  - Zambon Investigative Site, Frankfurt am Main
  - Zambon Investigative Site, Hamburg
  - Zambon Investigative Site, Hanover
  - Zambon Investigative Site, Lübeck
  - Zambon Investigative Site, München
  - Zambon Investigative Site, Münster
- Zambon Investigative Site, Athens, Greece
- Israel (6):
  - Zambon Investigative Site, Haifa
  - Zambon Investigative Site, Jerusalem
  - Zambon Investigative Site, Kfar Saba
  - Zambon Investigative Site, Petah Tikva
  - Zambon Investigative Site, Rehovot
  - Zambon Investigative Site, Ẕerifin
- Italy (10):
  - Zambon Investigative Site, Orbassano, TO
  - Zambon Investigative Site, Bari
  - Zambon Investigative Site, Brescia
  - Zambon Investigative Site, Foggia
  - Zambon Investigative Site, Milan
  - Zambon Investigative Site, Monza
  - Zambon Investigative Site, Palermo
  - Zambon Investigative Site, Pavia
  - Zambon Investigative Site, Pisa
  - Zambon Investigative Site, Roma
- Zambon Investigative Site, Groningen, Netherlands
- New Zealand (4):
  - Zambon Investigative Site, Auckland
  - Zambon Investigative Site, Christchurch
  - Zambon Investigative Site, Dunedin
  - Zambon Investigative Site, Hamilton West
- Portugal (8):
  - Zambon Investigative Site, Aveiro
  - Zambon Investigative Site, Braga
  - ZambonInvestigative Site, Coimbra
  - Zambon Investigative Site, Guimarães
  - Zambon Investigative site, Lisbon
  - Zambon Investigative Site, Loures
  - Zambon Investigative Site, Porto
  - Zambon Investigative Site, Vila Nova de Gaia
- Spain (9):
  - Zambon Investigative Site, A Coruña
  - Zambon Investigative Site, Barcelona
  - Zambon Investigative Site, Lleida
  - Zambon Investigative Site, Madrid
  - Zambon Investigative Site, Santander
  - Zambon Investigative Site, Seville
  - Zambon Investigative Site, Torrejón de Ardoz
  - Zambon Investigative Site, Usansolo
  - Zambon Investigative Site, Valencia
- Zambon Investigative Site, Sankt Gallen, Switzerland
- United Kingdom (13):
  - Zambon Investigative Site, Cambridge
  - Zambon Investigative Site, Cardiff
  - Zambon Investigative site, Dundee
  - Zambon Investigative Site, Edinburgh
  - Zambon Investigative Site, Gillingham
  - Zambon Investigative Site, Glasgow
  - Zambon Investigative Site, Kirkcaldy
  - Zambon Investigational site, Liverpool
  - Zambon Investigative Site, Llanelli
  - Zambon Investigative Site, London
  - Zambon investigative Site, Manchester
  - Zambon Investigative Site, Newcastle upon Tyne
  - Zambon Investigative Site, Worcester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was halted with 377 subjects randomised.
Groups:
- CMS (Colistimethate Sodium): Inhaled colistimethate sodium twice daily. The active pharmaceutical ingredient consisting of pure CMS one million international units (MIU) / 80 mg of CMS / 33 mg colistin base activity (CBA) was provided as a powder for nebuliser solution in 10R International Organization for Standardization (ISO) glass vials
  CMS: 1 M units equivalent to 80 mg colistimethate sodium diluted in 1 mL saline solution 0.45%. Investigational Medicinal Product (IMP) glass vials were shrink wrapped in opaque white plastic and provided in boxes of 30 vials (two weeks of b.i.d dosing).
  The 1 MIU/mL CMS/0.45% saline solution was transferred from the glass vial into a nebuliser system fitted with a 0.3 mL medication chamber, for administration by inhalation. This delivered a nominal dose of 0.3 MIU/24 mg CMS (~10 mg CBA) from the device.
  The first dose of the IMP was administered at the site under the supervision of the site staff and pts were instructed how to prepare and self-administer the IMP at home via the nebulizer system, b.i.d (morning and evening) over a period of 12 months.
  At least 10 minutes (min) before each administration, an inhaled short-acting bronchodilator (e.g., salbutamol /albuterol), supplied by the Sponsor, could be taken to improve tolerability.
- Placebo: Saline solution inhaled twice daily, provided and adminitered at the same way of the IMP.
  Placebo: 1 ml saline solution 0.45%. the placebo was made up of identical empty glass vials to which the same saline diluent was added in exactly the same way as the reconstitution of the active treatment by injecting the diluent through the rubber stopper. The glass vials were shrink wrapped with opaque white plastic to maintain the blind.
Period: Overall Study
Arm/Group | CMS (Colistimethate Sodium) | Placebo
Started | 177 | 200
Modified Intention to Treat Population - (mITT) | 176 | 197
Safety Population (SAF) | 176 | 197
Per -Protocol Population (PP) | 117 | 122
Completed | 123 | 129
Not Completed | 54 | 71
Not completed — Withdrawal by Subject | 32 | 27
Not completed — Adverse Event | 17 | 24
Not completed — Death | 0 | 1
Not completed — Non-Compliance with Study Drug | 1 | 0
Not completed — Protocol-Specified withdrawal criterion met | 3 | 16
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Population: The Intention-To-Treat Population will include all subjects who provided informed consent and received a patient number (randomisation number) whether or not they receive IMP.
Groups:
- CMS (Colistimethate Sodium): Inhaled colistimethate sodium twice daily. The active pharmaceutical ingredient consisting of pure CMS one million international units (MIU) / 80 mg of CMS / 33 mg colistin base activity (CBA) was provided as a powder for nebuliser solution in 10R International Organization for Standardization (ISO) glass vials
  CMS: 1 MIU equivalent to 80 mg colistimethate sodium diluted in 1 mL saline solution 0.45%. Investigational Medicinal Product (IMP) glass vials were shrink wrapped in opaque white plastic and provided in boxes of 30 vials (two weeks of b.i.d dosing).
  The 1 MIU/mL CMS/0.45% saline solution was transferred from the glass vial into a specific nebuliser system fitted with a 0.3 mL medication chamber, for administration by inhalation. This delivered a nominal dose of 0.3 MIU/24 mg CMS (~10 mg CBA) from the device.
  The first dose of the IMP was administered at the site under the supervision of the site staff and subjects were instructed how to prepare and self-administer the IMP at home via a specific nebuliser system, b.i.d (morning and evening) over a period of 12 months.
  At least 10 minutes (min) before each administration, an inhaled short-acting bronchodilator (e.g., salbutamol /albuterol), supplied by the Sponsor, could be taken to improve tolerability.
- Total: Total of all reporting groups
Arm/Group | CMS (Colistimethate Sodium) | Placebo | Total
Number analyzed (Participants) | 177 | 200 | 377
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 69 | 88 | 157
  >=65 years | 107 | 112 | 219
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age continuous data are provide for mITT Population that includes all subjects who provided informed consent, were randomised and received at least one dose or partial dose of study drug (summarised by randomised treatment)
  years
    number analyzed (Participants) | 176 | 197 | 373
    (all) | 64.2 (14.86) | 64.2 (13.06) | 64.2 (13.92)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex data are provide for mITT Population that includes all subjects who provided informed consent, were randomised and received at least one dose or partial dose of study drug (summarised by randomised treatment)
  Participants
    number analyzed (Participants) | 176 | 197 | 373
    Female | 123 | 126 | 249
    Male | 53 | 71 | 124
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity data are provide for mITT Population that includes all subjects who provided informed consent, were randomised and received at least one dose or partial dose of study drug (summarised by randomised treatment)
  Participants
    number analyzed (Participants) | 176 | 197 | 373
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 5 | 3 | 8
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 167 | 189 | 356
    More than one race | 0 | 1 | 1
    Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  Greece | 8 | 9 | 17
  New Zealand | 6 | 13 | 19
  Netherlands | 1 | 0 | 1
  Belgium | 0 | 2 | 2
  Italy | 23 | 30 | 53
  United Kingdom | 18 | 15 | 33
  Israel | 19 | 22 | 41
  Australia | 33 | 30 | 63
  Portugal | 21 | 27 | 48
  Switzerland | 1 | 0 | 1
  Germany | 32 | 33 | 65
  Spain | 15 | 19 | 34

OUTCOME MEASURES:

1. Primary Outcome: Mean Annual Non-cystic Fibrosis Bronchiectasis (NCFB) Pulmonary Exacerbation Rate
Description: The primary efficacy assessment for an individual subject was the frequency of pulmonary exacerbations (exacerbation rate). A pulmonary exacerbation was defined as the presence concurrently of at least three of the following eight symptoms/signs for at least 24 hours:
  * increased cough;
  * increased sputum volume and/or consistency;
  * increased sputum purulence;
  * new or increased haemoptysis;
  * increased wheezing;
  * increased dyspnoea;
  * increased fatigue/malaise;
  * episodes of fever (temperature ≥38°C). AND It was clinically determined that the subject required and was prescribed systemic antibiotic therapy. AND The episode of exacerbation lasted for at least 24 hours. The overall episode of exacerbation needs to last at least 24 hours, but individual symptoms/signs can last less than 24 hours (e.g, a temperature).
  AND in the opinion of the Investigator, the subject required and started treatment with systemic antibiotics.
Time Frame: 12 months
Population: The Modified ITT (mITT) Population will comprise all subjects who provided informed consent, were randomised and received at least 1 dose or partial dose of the IMP.
Measure: Least Squares Mean (95% Confidence Interval); unit: number of Pulmonary Exacerbations
Groups:
- CMS (Colistimethate Sodium): Inhaled colistimethate sodium twice daily. The active pharmaceutical ingredient consisting of pure CMS one million international units (MIU) / 80 mg of CMS / 33 mg colistin base activity (CBA) was provided as a powder for nebuliser solution in 10R International Organization for Standardization (ISO) glass vials.
  CMS: 1 MIU equivalent to 80 mg colistimethate sodium diluted in 1 mL saline solution 0.45%. Investigational Medicinal Product (IMP) glass vials were shrink wrapped in opaque white plastic and provided in boxes of 30 vials (two weeks of b.i.d dosing).
  The 1 MIU/mL CMS/0.45% saline solution was transferred from the glass vial into a specific nebuliser system fitted with a 0.3 mL medication chamber, for administration by inhalation. This delivered a nominal dose of 0.3 MIU/24 mg CMS (~10 mg CBA) from the device.
  The first dose of the IMP was administered at the site under the supervision of the site staff and subjects were instructed how to prepare and self-administer the IMP at home via a specific nebuliser system, b.i.d (morning and evening) over a period of 12 months.
  At least 10 minutes (min) before each administration, an inhaled short-acting bronchodilator (e.g., salbutamol /albuterol), supplied by the Sponsor, could be taken to improve tolerability.
Arm/Group | CMS (Colistimethate Sodium) | Placebo
Number analyzed (Participants) | 176 | 197
number of Pulmonary Exacerbations | 0.580 [NA to NA] — The CIs of the LS Mean NCFB pulmonary exacerbation annual rates are infinite in both the CMS and placebo groups due to the SEs being not-estimable. (the low numbers of subjects and/or events in some countries led to the LS Means being not-estimable). | 0.948 [NA to NA] — The CIs of the LS Mean NCFB pulmonary exacerbation annual rates are infinite in both the CMS and placebo groups due to the SEs being not-estimable. (the low numbers of subjects and/or events in some countries led to the LS Means being not-estimable).
Statistical Analysis 1: Comparison: CMS (Colistimethate Sodium) vs Placebo; Test type: Superiority — The number of NCFB pulmonary exacerbations was compared between treatment groups using a negative binomial model including treatment, pooled site (country) and baseline use of stable concomitant therapy with oral macrolides as fixed effects and log-time on treatment as an offset; p = 0.00101, two-sided Wald chi-square test; LS Mean rate ratio = 0.612, 95% CI 2-sided [0.457 to 0.820]

ADVERSE EVENTS:
Time Frame: All AEs occurring from the day of the first IMP administration, i.e. Visit 2 (day 0), up to the follow-up (54 weeks after the beginning of the trial), when follow-up phone call took place.
Description: An AE is "any untoward medical occurrence in a patient or clinical trial subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment". An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an IMP, whether or not considered related to the IMP.
Groups:
- CMS (Colistimethate Sodium) (SAF): Inhaled colistimethate sodium twice daily. The active pharmaceutical ingredient consisting of pure CMS one million international units (MIU) / 80 mg of CMS / 33 mg colistin base activity (CBA) was provided as a powder for nebuliser solution in 10R International Organization for Standardization (ISO) glass vials.
  CMS: 1 MIU equivalent to 80 mg colistimethate sodium diluted in 1 mL saline solution 0.45%. Investigational Medicinal Product (IMP) glass vials were shrink wrapped in opaque white plastic and provided in boxes of 30 vials (two weeks of b.i.d dosing).
  The 1 MIU/mL CMS/0.45% saline solution was transferred from the glass vial into a specific nebulizer system fitted with a 0.3 mL medication chamber, for administration by inhalation. This delivered a nominal dose of 0.3 MIU/24 mg CMS (~10 mg CBA) from the device.
  The first dose of the IMP was administered at the site under the supervision of the site staff and subjects were instructed how to prepare and self-administer the IMP at home via a specific nebulizer system, b.i.d (morning and evening) over a period of 12 months.
  At least 10 minutes (min) before each administration, an inhaled short-acting bronchodilator (e.g., salbutamol /albuterol), supplied by the Sponsor, could be taken to improve tolerability.
- Placebo (SAF): Saline solution inhaled twice daily, provided and administered at the same way of the IMP.
  Placebo: 1 ml saline solution 0.45%. The placebo was made up of identical empty glass vials to which the same saline diluent was added in exactly the same way as the reconstitution of the active treatment by injecting the diluent through the rubber stopper. The glass vials were shrink wrapped with opaque white plastic to maintain the blind.
Arm/Group | CMS (Colistimethate Sodium) (SAF) | Placebo (SAF)
All-Cause Mortality (participants affected / at risk) | 1/176 | 1/197
Serious Adverse Events (participants affected / at risk) | 31/176 | 46/197
Other Adverse Events (participants affected / at risk) | 142/176 | 159/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CMS (Colistimethate Sodium) (SAF) (N=176) | Placebo (SAF) (N=197)
Infective exacerbation of bronchiectasis (Infections and infestations) | 15 (17) | 29 (36)
Pneumonia (Infections and infestations) | 4 (4) | 5 (5)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Extradural abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Spinal cord infection (Infections and infestations) | 1 (1) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CMS (Colistimethate Sodium) (SAF) (N=176) | Placebo (SAF) (N=197)
Infective exacerbation of bronchiectasis (Infections and infestations) | 67 (110) | 110 (196)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (24) | 19 (19)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 (34) | 16 (19)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 9 (19) | 19 (33)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 7 (9)
Diarrhoea (Gastrointestinal disorders) | 12 (12) | 5 (5)
Headache (Nervous system disorders) | 4 (4) | 11 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/74/NCT03093974/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/74/NCT03093974/SAP_001.pdf